CLINICAL TRIAL: NCT02143622
Title: A Phase Ib/II, Multicenter Study of LJM716 in Combination With Cetuximab in Patients With Platinum-pretreated Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Study of Efficacy and Safety of LJM716 and Cetuximab in Head and Neck Squamous Cell Carcinoma Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLJM716X2104
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — elgemtumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LJM716+cetuximab (Experimental)
  Interventions: Biological: LJM716; Biological: cetuximab

INTERVENTIONS:
Biological: LJM716 — antibody
Biological: cetuximab — antibody

SUMMARY:
To establish whether LJM716 in combination with cetuximab is safe and has beneficial effects in patients with platinum-pretreated recurrent/metastatic head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Most recent regimen contains both platinum and cetuximab (Phase II, group B).
* ECOG Performance Status (PS) ≤ 2.
* Recovery from all AEs of previous anti-cancer therapies, to baseline or to CTCAE Grade ≤ 1, except for alopecia.
* Measurable disease as determined by RECIST v1.1.

Exclusion Criteria:

* Previous anti-HER3 antibody treatment.
* Symptomatic brain metastasis.
* Prior systemic anti-cancer treatment, within a period of time that is shorter than the cycle length used for that treatment prior to starting study treatment.
* Prior anaphylactic or other severe infusion reaction to human immunoglobulin or antibody formulations.
* Inadequate end organ function.
* Ongoing diarrhea CTCAE Grade ≥ 2. Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Target lesion change compared to baseline in patients, per RECIST 1.1 | 6 months
  Assessment of the preliminary anti-tumor activity of LJM716 in combination. Change in target lesion measurements, from baseline as per RECIST 1.1
Phase Ib: Number of Total Dose-limiting Toxicity (DLT) During Dose Escalation to Determine Maximum Tolerated Dose (MTD) | 35 days
  The dose escalation part of the study will be guided by a well-established statistical method/model to estimate the maximum tolerated dose of LJM716 in combination with cetuximab
Phase II: Percentage of Patients with an Objective Overall Response (OOR) per RECIST 1.1 | 6 months
  Patients with an Objective Overall Response (OOR) were those whose best response to treatment was a complete response (CR) or a partial response (PR) assessed by imaging, as pr RECIST 1.1.

SECONDARY OUTCOMES:
Safety and tolerability of the LJM716- cetuximab combination | 6 months
  This will be assessed by looking at the number of Adverse Events (AEs), serious AEs (SAEs) changes in hematology and chemistry values, vital signs, electrocardiograms (ECGs), dose interruptions, reductions and dose intensity.
blood concentration versus time profiles blood PK parameters of LJM716 and cetuximab concentration | 6 months
  blood concentration versus time profiles blood PK parameters will be used to characterize the PK profiles of LJM716 and cetuximab concentration when used in combination
Best overall response (BOR), per RECIST 1.1 | 6 months
  BOR will be used to further assess the anti-tumor activity of LJM716-cetuximab combination.
Duration of response (DOR) per RECIST 1.1 | 6 months
  Duration of response will be used to further assess the anti-tumor activity of LJM716-cetuximab combination
Overall survival (OS) per RECIST 1.1 | 12 months
  Overall survival will be used to further assess the anti-tumor activity of LJM716-cetuximab combination
Progression free survival (PFS) per RECIST 1.1 | 6 months
  Progression free survival will be used to further assess the anti-tumor activity of LJM716-cetuximab combination

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals